CLINICAL TRIAL: NCT00106782
Title: Placebo Controlled Study of the Therapeutic Effect of the Transcranial Electrical Polarization in Patients With Focal Hand Dystonia
Brief Title: Transcranial Electrical Polarization to Treat Focal Hand Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Mark Hallett, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050122; 05-N-0122
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-14

CONDITIONS: Dystonia; Focal Hand Dystonia; FHD
Keywords: Electrical; Stimulation; Dystonia; Brain; Focal Hand Dystonia; FHD
MeSH Terms: conditions — Dystonia; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 1 (Other): Real TEP
  Interventions: Procedure: Transcranial Electrical Polarization (TEP)
- 2 (Other): Sham Stimulation
  Interventions: Procedure: Transcranial Electrical Polarization (TEP)

INTERVENTIONS:
Procedure: Transcranial Electrical Polarization (TEP)

SUMMARY:
This study will evaluate the effect of transcranial electrical polarization (TEP), also called direct current (DC) stimulation, on focal hand dystonia in people with writer's cramp. In dystonia, muscle spasms cause uncontrolled twisting and repetitive movement or abnormal postures. Focal dystonia involves just one part of the body, such as the hand, neck or face. When people with focal hand dystonia make small and repeated movements with their hands, there is extra activity in the part of the brain called the motor cortex. TEP is a method of brain stimulation that slows down the activity of the nerve cells in the motor cortex. This study may help researchers develop new ways to treat focal hand dystonia.

People 18 years of age and older with focal hand dystonia may be eligible for this study. Participants have a neurological examination and are randomly assigned to one of two treatment groups: TEP or placebo stimulation. The TEP group receives stimulation to the parts of the brain used for hand movement, and the placebo group receives sham stimulation, which does not affect any area of the brain. There are three TEP/placebo sessions over a period of 7 to 10 days. The first session may last up to 2-1/2 hours; the other two sessions last 1-2 hours.

For TEP, sponge electrodes are placed on the scalp and an electrical current is passed through the scalp and skull to the outer part of brain. Before and after each session, participants have a neurological examination, including an evaluation of the rate and severity of their movement problems. For this assessment, participants do a writing test while the electrical activity of their hand muscles is recorded using surface electromyography (EMG). For EMG, small metal disks (electrodes) filled with a conductive gel are taped to the skin over the muscles being tested.

Patients are followed in the clinic the day after the end of TEP treatment for evaluation of their movement abilities and the effects of therapy, such as improvement of handwriting.

DETAILED DESCRIPTION:
Objective: The treatment of focal hand dystonia (FHD) needs further improvement. A deficiency of inhibition was demonstrated in patients with writer's cramp. The passage of weak DC currents across the head, or transcranial electrical polarization (TEP) has been done for many years with numerous effects described in healthy subjects and mentally diseased patients. Recently, it has been shown by objective means, in controlled experiments, that this type of treatment has robust and lasting effects on the excitability of the motor cortex in healthy humans.

Study population: 40 subjects with focal hand dystonia.

Design: We hypothesize that TEP will have a beneficial effect on hand writing in patients with FHD because it will decrease the excitability of the motor cortex compensating the deficiency of inhibition. Specifically, we propose to look at the effect of 2 mA TEP with cathode position over the hand projection in the contralateral to the affected hand primary motor cortex. Anodes will be placed over the orbit and mastoid process ipsilateral to the affected hand (contralateral to the cathode). Over a two-year period, we will enroll 40 patients with FHD and evaluate the acute TEP effects over a period of 1 week (3 TEP sessions).

Outcome measures: Symptoms will be evaluated by kinematic analysis of the handwriting and with dystonia scales.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with focal hand dystonia 18 years old or older will be included.

EXCLUSION CRITERIA:

Exclusion criteria will include the standard exclusions for TEP as well as exclusions specific to this study.

We will exclude subjects with:

* Any significant medical or psychiatric illness (other than FHD).
* Patients with a positive pregnancy test will be excluded because the effects of TEP on the fetus is unknown. A urine sample for pregnancy testing will be obtained prior to the TEP, and on the day of the first TEP session.
* History of epilepsy.
* Concurrent use of neuroleptic agents.
* Any other licit or illicit drugs other that could lower the seizure threshold.
* Metal implants.
* Who have received botulinum toxin injection within 10 weeks of starting the protocol.
* Secondary hand dystonia.
* Mentally impaired patients having no capacity to provide their own consent will be excluded from the study because such patients may have difficulty performing the required test.
* If participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as excessive fatigue, general frailty, or excessive apprehension.
* Unable or unwilling to refrain from alcohol for 24 hours prior to study days.

Patients may continue taking muscle relaxants, artane and other anticholinergic drugs, L-DOPA and dopamine agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-03-18; Primary Completion 2010-05-14 (Actual); Study Completion 2010-05-14 (Actual)

PRIMARY OUTCOMES:
The Fahn Dystonia Scale before and after real and placebo TEP course. | 1 week post-TEP

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agnew WF, McCreery DB. Considerations for safety in the use of extracranial stimulation for motor evoked potentials. Neurosurgery. 1987 Jan;20(1):143-7. doi: 10.1097/00006123-198701000-00030. PMID 3808255
- [Background] Antal A, Nitsche MA, Paulus W. External modulation of visual perception in humans. Neuroreport. 2001 Nov 16;12(16):3553-5. doi: 10.1097/00001756-200111160-00036. PMID 11733710
- [Background] Chen R, Wassermann EM, Canos M, Hallett M. Impaired inhibition in writer's cramp during voluntary muscle activation. Neurology. 1997 Oct;49(4):1054-9. doi: 10.1212/wnl.49.4.1054. PMID 9339689